CLINICAL TRIAL: NCT04606524
Title: Relationship Between MUC1 Expression and Gustatory Function in Postmenopausal Females
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amira Abdelwhab, Dr., October 6 University
Other Study IDs: 8-2020
Record Dates: First submitted 2020-08-29; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Taste, Altered
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Analysis of epithelial oral mucosal MUC1 expression level in saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- study group: 25 postmenopausal females will be included in this study
- control group: 25 premenopausal females will be included in this tudy

SUMMARY:
50 females will be included in this study. they will be divided into 2 groups (study group which will include 25 postmenopausal females - and control group which will include premenopausal females) For testing gustatory function, a whole mouth above threshold taste test will be carried out in which a concentration of sucrose, sodium chloride, citric acid and quinine hydrochloride solutions were used for sweet, salty, sour and bitter types of taste respectively .

Saliva will be collected to evaluate MUC1 expression

DETAILED DESCRIPTION:
50 females will be included in this study. they will be divided into 2 groups (study group which will include 25 postmenopausal females - and control group which will include premenopausal females)

For testing gustatory function, a whole mouth above threshold taste test will be carried out in which a concentration of sucrose, sodium chloride, citric acid and quinine hydrochloride solutions were used for sweet, salty, sour and bitter types of taste respectively . Five concentration levels (in ½ log steps) of sodium chloride (0.01-1.0 mM), citric acid (0.32-0.032 mol l-1), quinine hydrochloride (0.01- 1.0 mM) and sucrose (0.01-1.0 mM) will be prepared in 5 ml samples. All the solutions will be made with distilled water. The intensity threshold of taste perception of each solution will be determined by scoring the lowest concentration as 5' and the highest concentration as 1'. The solutions will be given in increasing concentrations. The patient then should identify the quality (salty, sour, sweet, bitter or tasteless) and intensity of each test solution . Quality judgments for each solution will be coded as correct, incorrect or tasteless by asking subjects to name the taste they perceived.

Saliva will be collected in the morning between 9:00 am and 11:00 am. Patient will be instructed to stop eating and drinking at least 2 h before sample collection. Chewing 1 g of gum base will be used to stimulate salivary flow. The saliva that will be collected for the first 2 min will be discarded, and then Stimulated whole saliva will be collected for the next 10 min with the mechanical chewing stimulation.

Two milliliters of Stimulated whole saliva from each participant will be collected and added to RNA stabilizing solution and used for RNA extraction. The SWS samples will be centrifuged at 10,000 g for 20 min at 48C to remove any cellular debris. The clarified supernatants will be aliquoted and frozen at 70 C for analytic experiments.

this is to determination of oral mucosal epithelial MUC1 expression level

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for study group include individuals who are in the age range of 50-75 years, history of complete amenorrhoea patients who are not taking any medication [including hormone replacement therapy (HRT) for female patients]. Also females who are not a denture wearer and those who are having good oral hygiene.

Inclusion criteria for study group include individuals who are in the range between 20-40 years with normal menstrual cycle of 28 to 30 days. they should be healthy volunteers free from any systemic diseases

Exclusion Criteria:

* Exclusion criteria for both groups include patients having any oral diseases (like oral candidiasis)
* those who have any systemic diseases (such as diabetes, nutritional deﬁciency, cardiovascular, respiratory and endocrinal disorders).
* Also any history that could aﬀect gustatory function (e.g medications &radiotherapy or smoking

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: study will include 50 healthy females free from any systemic diseases or inder any medications that may affect gustatory function divided into 2 groups study group and it will include 25 postmenopausal females control group it will include 25 postmenopausal females
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Alterations of the gustatory function in postmenopausal females | 12-18 month
  , a whole mouth above threshold taste test will be carried out in which a concentration of sucrose, sodium chloride, citric acid and quinine hydrochloride solutions were used for sweet, salty, sour and bitter types of taste respectively

SECONDARY OUTCOMES:
MUC1 expression | 12-18 month
  Two milliliters of Stimulated whole saliva from each participant will be collected and added to RNA stabilizing solution and used for RNA extraction

CONTACTS AND LOCATIONS:
Overall Officials: reham aggour, Study Director — October 6 University

IPD SHARING:
Plan to Share IPD: Undecided